CLINICAL TRIAL: NCT06544655
Title: A Phase 1/1b First-in-human Trial of BMS-986484 as Monotherapy and Combination Therapy in Participants With Advanced Solid Malignancies
Brief Title: A Study of BMS-986484 Alone and Combination Therapy in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA233-0000; EU 2024-513696-40 (Registry Identifier: EU Trial Number)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors
Keywords: Opdivo®; Immunotherapy; BMS-986484; Non-small cell lung cancer (NSCLC); Microsatellite stable (MSS) colorectal carcinoma (CRC); Pancreatic ductal adenocarcinoma (PDAC); Gastric/gastroesophageal junction adenocarcinoma (G/GEJC); Squamous cell carcinoma of the head and neck (SCCHN); anti-CD40; anti-FAP; FOLFOX; CAPOX; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Spinocerebellar Degenerations; Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Nivolumab; Oxaliplatin; Capecitabine; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1A: BMS-986484 Dose Escalation (Experimental)
  Interventions: Drug: BMS-986484
- Part 1B: BMS-986484 + Nivolumab Dose Escalation (Experimental)
  Interventions: Drug: BMS-986484; Biological: Nivolumab
- Part 2A: BMS-986484 Dose Expansion (Experimental)
  Interventions: Drug: BMS-986484
- Part 2B: BMS-986484 + Nivolumab Dose Expansion (Experimental)
  Interventions: Drug: BMS-986484; Biological: Nivolumab
- Part 1C: BMS-986484 + Nivolumab + Chemotherapy Dose Escalation (Experimental)
  Interventions: Drug: BMS-986484; Biological: Nivolumab; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Fluorouracil; Drug: Calcium folinate
- Part 1 Co-Admin: BMS-986484 + Nivolumab (Experimental)
  Interventions: Drug: BMS-986484; Biological: Nivolumab
- Part 1SC: BMS-986484 Monotherapy Subcutaneous Dose Escalation (Experimental)
  Interventions: Drug: BMS-986484
- Part 2C: BMS-986484 + Nivolumab + Chemotherapy Dose Expansion (Experimental)
  Interventions: Drug: BMS-986484; Biological: Nivolumab; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Fluorouracil; Drug: Calcium folinate

INTERVENTIONS:
Drug: BMS-986484 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
  Arms: Part 1 Co-Admin: BMS-986484 + Nivolumab; Part 1B: BMS-986484 + Nivolumab Dose Escalation; Part 1C: BMS-986484 + Nivolumab + Chemotherapy Dose Escalation; Part 2B: BMS-986484 + Nivolumab Dose Expansion; Part 2C: BMS-986484 + Nivolumab + Chemotherapy Dose Expansion
Drug: Oxaliplatin — Specified dose on specified days
  Arms: Part 1C: BMS-986484 + Nivolumab + Chemotherapy Dose Escalation; Part 2C: BMS-986484 + Nivolumab + Chemotherapy Dose Expansion
Drug: Capecitabine — Specified dose on specified days
  Arms: Part 1C: BMS-986484 + Nivolumab + Chemotherapy Dose Escalation; Part 2C: BMS-986484 + Nivolumab + Chemotherapy Dose Expansion
Drug: Fluorouracil — Specified dose on specified days
  Arms: Part 1C: BMS-986484 + Nivolumab + Chemotherapy Dose Escalation; Part 2C: BMS-986484 + Nivolumab + Chemotherapy Dose Expansion
Drug: Calcium folinate — Specified dose on specified days
  Arms: Part 1C: BMS-986484 + Nivolumab + Chemotherapy Dose Escalation; Part 2C: BMS-986484 + Nivolumab + Chemotherapy Dose Expansion

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMS-986484 administered alone, in combination with nivolumab in participants with advanced/metastatic solid tumors including non-small cell lung cancer (NSCLC), microsatellite stable (MSS) colorectal carcinoma (CRC), pancreatic ductal adenocarcinoma (PDAC), gastric/gastroesophageal junction adenocarcinoma (G/GEJC), and squamous cell carcinoma of the head and neck (SCCHN).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced unresectable, metastatic, or recurrent malignant tumors including non-small cell lung cancer (NSCLC), pancreatic ductal adenocarcinoma (PDAC), gastric/gastroesophageal junction adenocarcinoma (G/GEJC), microsatellite stable colorectal cancer (MSS CRC), and squamous cell carcinoma of the head and neck (SCCHN).
* Must have measurable disease by response evaluation criteria in solid tumors version 1.1 (RECIST v1.1).
* Must have an Eastern Cooperative Oncology Group Performance Status of 0 or 1.

Exclusion Criteria:

* History of or with active interstitial lung disease or pulmonary fibrosis.
* Active, known, or suspected autoimmune disease.
* Serious uncontrolled medical disorders.
* New onset, non-catheter-associated venous thromboembolism within the past 6 months.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-10-14 (Estimated); Study Completion 2027-10-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to approximately 2 years
Incidence of serious adverse events (SAEs) | Up to approximately 2 years
Incidence of AEs meeting protocol defined dose-limiting toxicity (DLT) criteria | Up to approximately 28 days
Incidence of AEs leading to discontinuation | Up to approximately 2 years
Incidence of AEs leading to death | Up to approximately 2 years

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to approximately 2 years
Time of maximum observed concentration (Tmax) | Up to approximately 2 years
Area under the concentration-time curve (AUC) | Up to approximately 2 years
Incidence of anti-drug antibodies (ADAs) | Up to approximately 2 years
Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | Up to approximately 2 years
Disease control rate (DCR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | Up to approximately 2 years
Duration of response (DOR) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- United States (5):
  - University of Arizona Cancer Center, Tucson, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - START Midwest, Grand Rapids, Michigan
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - NEXT Oncology, San Antonio, Texas
- Australia (2):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
- Japan (2):
  - Local Institution - 0023, Chuo-ku, Tokyo
  - Local Institution - 0022, Kashiwa

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06544655.html